CLINICAL TRIAL: NCT05772676
Title: The Effect of Aprepitant Reducing Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Gastric Sleeve Surgery
Brief Title: The Effect of Aprepitant Reducing Postoperative Nausea and Vomiting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital General Tlahuac (Other Government)
Responsible Party: Principal Investigator, CARLOS ZERRWECK LOPEZ, Professor of Surgery, UNAM, Hospital General Tlahuac
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: APREPITANTBAJAMED-01-2023
Record Dates: First submitted 2023-02-09; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Nausea and Vomiting, Postoperative
Keywords: Laparoscopic Gastric Sleeve; Bariatric Surgery; Nausea and Vomiting, Postoperative; Aprepitant
MeSH Terms: conditions — Obesity; Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial conducted in obese patients undergoing laparoscopic gastric sleeve surgery to assess the efficacy of Aprepitant (80 or 125 mg) in combination with a standard antiemetic regimen (Ondansetron + Metoclopramide + Dexamethasone) is presented vs placebo + the same standard regimen, evaluating postoperative nausea and vomiting by means of a specific scale (Rhodes index) for the assessment of nausea and vomiting
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple-blinded, 1:1ratio to Aprepitant or placebo
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aprepitant (Experimental): Aprepitant (80 or 125 mg) + Ondansetron 8 mg + Metoclopramide 10 mg + Dexamethasone 8 mg
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Placebo + Ondansetron 8 mg + Metoclopramide 10 mg + Dexamethasone 8 mg
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aprepitant — 80 or 125 mg tablet + standard antiemetic regimen, once two hours before surgery
  Arms: Aprepitant
Other: Placebo — Placebo + standard antiemetic regimen, once two hours before surgery
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of Aprepitant + standard antiemetic regimen in reducing postoperative nausea and vomiting after laparoscopic gastric sleeve versus placebo + standard antiemetic regimen

DETAILED DESCRIPTION:
After being informed about the study, all patients who provide written informed consent and meet the eligibility requirements will be randomized in a triple-blind manner (participant, evaluator, and investigator) in a 1:1 ratio to Aprepitant (80 or 125 mg) + standard antiemetic regimen (once two hours before surgery) or placebo + standard antiemetic regimen(once two hours before surgery).

The standard antiemetic regimen will be Ondansetron 8 mg + Metoclopramide 10 mg + Dexamethasone 8 mg

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old.
* Non-smokers.
* Obesity with BMI > 30 kg/m2.
* Undergoing laparoscopic gastric sleeve.

Exclusion Criteria:

* Documented hypersensitivity to any component of the study regimen.
* Current treatment with: Orap (pimozide), Seldane (terfenadine), Hismanal (astemizole) or Propulsid (cisapride).
* Allergy to opioid drugs used in the anesthetic protocol.
* Drug or alcohol abuse.
* Chronic nausea and vomiting.
* Previous bariatric procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient's postoperative nausea and vomiting evaluation at 0 hrs (Rhodes index) | 0 postoperative hours
  Change of postoperative nausea and vomiting after laparoscopic gastric sleeve using Rhodes scale
Patient's postoperative nausea and vomiting evaluation at 6 hrs (Rhodes index) | 6 postoperative hours
  Change of postoperative nausea and vomiting after laparoscopic gastric sleeve using Rhoades scale
Patient's postoperative nausea and vomiting evaluation at 12 hrs (Rhodes index) | 12 postoperative hours
  Change of postoperative nausea and vomiting after laparoscopic gastric sleeve using Rhoades scale
Patient's postoperative nausea and vomiting evaluation at 24 hrs (Rhodes index) | 24 postoperative hours
  Change of postoperative nausea and vomiting after laparoscopic gastric sleeve using Rhoades scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Tlahuac, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No